CLINICAL TRIAL: NCT03081897
Title: Influence of Regional Anaesthesia on the Expression of Substance P During Unilateral Neck Dissection Due to Head and Neck Cancer
Brief Title: Regional Anaesthesia and Substance P in Head and Neck Cancer
Acronym: SPRANC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: for organizational reasons
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jurgen Birnbaum, Principal Investigator of the Department of Anesthesiology and Intensive Care Medicine, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA1/119/16
Record Dates: First submitted 2016-07-28; First posted 2017-03-16 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPRANC Block group (Experimental): General anaesthesia and additional regional anaesthesia (cervical plexus block) on the tumor side.
  Interventions: Drug: SPRANC Block group
- SPRANC Control group (Active Comparator): General anaesthesia
  Interventions: Drug: SPRANC Control group

INTERVENTIONS:
Drug: SPRANC Block group — General anaesthesia with Propofol (2mg/kgKG) and Remifentanil (0,1-0,4 µg/kg/min); additional regional anaesthesia (cervical plexus block) with an long acting local anesthetic according to clinical estimation of the treating anesthetist (about 15 ml Ropivacaine 0,75% around the carotid bifurcation, 5 ml Ropivacaine in the region of Erb´s Point of the superficial cervical plexus and 10 ml Ropivacaine at the area of skin incision on the tumor side); unilateral neck dissection.
  Arms: SPRANC Block group
Drug: SPRANC Control group — General anaesthesia with Propofol (2mg/kgKG) and Remifentanil (0,1-0,4 µg/kg/min); additional regional Patient Control Group (no Intervention planned), general anaesthesia with Propofol (2mg/kgKG) and Remifentanil (0,1-0,4 µg/kg/min); unilateral neck dissection.
  Arms: SPRANC Control group

SUMMARY:
In the clinical trial the investigators will observe the impact of regional anesthesia in addition to a general anesthesia on the expression of substance P in patients with unilateral Head or Neck cancer undergoing unilateral Neck Dissection. The investigators will perform an unilateral regional cervical plexus block on the tumor side. The tissue of the tumor side will be analysed by immunohistology, measuring the expression of the Substance P.

DETAILED DESCRIPTION:
Several investigations show that anesthetic procedures, and especially the perioperative regional anesthesia, can have a benefit for patients undergoing tumor surgery.The perioperative regional anesthesia might reduce the immunological response and therefore lower the risk of tumor relapse. Factors that might play a role in tumor relapse are various, so more prospective and randomised trials are necessary to investigate the underlying mechanisms.

In a retrospective analysis by Merquiol et al. it was shown that an cervical epidural anesthesia was associated with an extended tumorfree timeline of larynx and hypopharynx carcinoma.

Supporting results could be seen in a study by Munoz et al. performing regional anaesthesia in breast cancer patients.

Taking all these facts into consideration the investigators believe that performing regional aneasthesia could reduce the relapse of larynx carcinoma. The relapse of carcinoma is believed to be linked to substance P and the neurokinin 1 (NK-1) receptor .

It is accepted that an additional regional anesthesia could reduce the impact of substance P to gain a normal immune response in the perioperative setting and to reduce the rate of tumor relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Charité - Universitaetsmedizin Berlin, Campus Charité Mitte
* Primary diagnosis of unilateral head or neck cancer
* Resection of Tumor is planned with unilateral neck dissection
* Patient did not underwent any therapeutic treatment of the cancer before start of study
* Surgical therapy is planned with curative intent

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulation disorders, which can lead to complications in regional anesthesia
* Insulin-dependent diabetes mellitus, polyneuropathy
* Severe psychiatric disorders
* Dementia
* Alcohol abuse, Korsakoff syndrome
* Medication with immunosuppressants or immune modulantia
* Patient under Special Care
* Refusal of study participation
* Pregnancy and breast feeding period.
* Participation in a clinical intervention study, parallel with the study or participation up to 30 days before inclusion
* Lack of consent that pseudonomized data of the study may be saved and distributed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Expression of Substance P | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Birnbaum, PD Dr, Principal Investigator — Charité Universiteaetsmedizin Berlin, Klinik fuer Anaesthesiologie, Campus Mitte
Locations (1):
- Charité Universitaetsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided